CLINICAL TRIAL: NCT02742870
Title: Diffusion Magnetic Resonance Imaging Using ADC (Apparent Diffusion Coefficient) Histograms in the Evaluation of Adnexal Tumor Aggressiveness
Brief Title: Diffusion MRI (Magnetic Resonance Imaging) Using ADC (Apparent Diffusion Coefficient) Histograms in the Evaluation of Adnexal Tumor Aggressiveness
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Mieke Cannie, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-MRI-Adnexal Tumor
Record Dates: First submitted 2016-04-01; First posted 2016-04-19 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Adnexal Tumor
Keywords: Diffusion MRI; ADC histograms; Adnexal tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with MRI pelvic imaging: Women over 18 years old, having undergone a magnetic resonance imaging of the pelvis within the CHU Brugmann Hospital
  Interventions: Other: Correlation of MRI results with clinical characteristics of the adnexal mass

INTERVENTIONS:
Other: Correlation of MRI results with clinical characteristics of the adnexal mass — Quantitative analysis of the magnetic resonance images realised with the Ingenia 3 Tesla Engine (Philips) and the Area 1,5 Tesla Engine (Siemens), based on the ADC cartography.The post-processing will be realized with the Syngo Onco Care application of Siemens, that allows an histogram analysis of the ADC of all sections of the adnexal mass, as opposed to a section per section approach with the Region of Interest (ROI) method.
  The results will be correlated with the clinical data regarding the adnexal mass: anatomo-pathology status (malignancy and aggressiveness of the tumor) and the gynecological follow-up.

SUMMARY:
Diffusion-weighted sequences have been routinely performed for years to study the pelvis. They have been so far mainly qualitatively interpreted, that is to say as the absence or presence of an hypersignal at a high b value. The quantitative analysis involves placing the region of interest (ROI) on the apparent diffusion coefficient (ADC) map. The manual placement is very operator dependent, and does not reflect the entirety of the studied mass.

In all fields of Magnetic Resonance Imaging, a multiparametric approach integrating diffusion analysis is flourishing. However, the quantitative analysis of the diffusion is still little studied for tumor heterogeneity analysis, including in the gynecological sphere.

The investigators will therefore retrospectively evaluate the apparent diffusion coefficient (ADC) histograms, extracted from the diffusion ponderation sequences, of the magnetic imaging resonance analysis of adnexal masses and confront the results with the anatomo-pathology results, for patients having undergone surgery, and/or with the clinical and imagery follow-up results.

The investigators goal will be to improve the performance of conventional MRI in the analysis of adnexal masses.

The expected benefits of this study are:

* a correlation with the histology analysis or the clinical monitoring
* an improved prediction of the malignancy of the tumor
* an improved magnetic resonance imaging performance for adnexal masses, with better surgical therapeutic management
* an improved negative predictive value, thereby ultimately limiting unnecessary surgical explorations.

ELIGIBILITY:
Inclusion Criteria:

- Women aged over 18 years old, having undergone magnetic resonance imaging of the pelvis within the CHU Brugmann hospital.

Exclusion Criteria:

* Examinations without diffusion sequences
* Examinations with incomplete diffusion sequences
* Absence of anato-pathologic result, or absence of gynecological clinical/imaging follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women having undergone magnetic resonance imaging of the pelvis within the CHU Brugmann hospital.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Apparent diffusion coefficient (ADC) of the adnexal mass volume (mm2/sec) | From 01/01/2015 till the end of study (2 years)
  Apparent diffusion coefficient (ADC) expressed in mm2/sec. Magnetic resonance images realised with the Ingenia 3 Tesla Engine (Philips) and the Area 1,5 Tesla Engine (Siemens).Post-processing realized with the Syngo Onco Care application of Siemens.
Anatomo-pathology classification - histological type | From 01/01/2015 till the end of study (2 years)
  Follow-up of the patients that did undergo surgery: histological type of tumor. The histological type of the tumor will be determined by the Anatomo-Pathology Department of the CHU Brugmann hospital, according to standard of care.
MRI Adnex score | From 01/01/2015 till the end of study (2 years)
  Follow-up of the patients that did not undergo surgery: medical imaging classification of the adnexal mass (MRI Adnex score)
IOTA ultrasound classification | From 01/01/2015 till the end of study (2 years)
  Follow-up of the patients that did not undergo surgery: transvaginal ultrasound classification of the adnexal masse (IOTA ultrasound classification)
Anatomo-pathology classification - malignancy grading of tumor | From 01/01/2015 till the end of study (2 years)
  Follow-up of the patients that did undergo surgery: malignancy grading of the adnexal mass according to FIGO classification.

CONTACTS AND LOCATIONS:
Overall Officials: Mieke Cannie, MD, Principal Investigator — CHU Brugmann; Nathalie Hottat, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Thomassin-Naggara I, Aubert E, Rockall A, Jalaguier-Coudray A, Rouzier R, Darai E, Bazot M. Adnexal masses: development and preliminary validation of an MR imaging scoring system. Radiology. 2013 May;267(2):432-43. doi: 10.1148/radiol.13121161. Epub 2013 Mar 6. PMID 23468574
- [Background] Just N. Improving tumour heterogeneity MRI assessment with histograms. Br J Cancer. 2014 Dec 9;111(12):2205-13. doi: 10.1038/bjc.2014.512. Epub 2014 Sep 30. PMID 25268373